CLINICAL TRIAL: NCT04806152
Title: Effect of Exercise on Muscle Mass, Functional Capacity and Physical Activity in Community-dwelling Elderly With Sarcopenia in Jamaica
Brief Title: Sarcopenia and Combined-modality Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID19 outbreak began March 2020 in Jamaica. Associated risks, prohibitive cost of mitigating those risks for study participants and locally enacted legislation militated against further recruitment and intervention activities.
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UWIJAMSarc
Record Dates: First submitted 2021-03-09; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia
Keywords: exercise; training
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenia and combined-modality high intensity supervised exercise training (Experimental): Participants were given Treadmill exercise training, lower extremity progressive resistance training using a Cybex leg press machine, and a 1-hour adaptive physical activity (APA) programme in which participants were required to walk for 12 minutes through an obstacle course in which they must clear 10 cm high boards, climb 3 steps and walk sideways through hula-hoops placed on the floor all the while dual-tasking i.e. waving at strategically placed signs, conversing while walking and picking up objects. Participants also performed exercises at the parallel bars which included weight-shifting from leg to leg and half-squatting; they were also guided through seated upper- and lower-limb stretching exercises for range of motion and trunk mobility. All exercise sessions were supervised by physiotherapists. For two of the weekdays on which participants did not attend supervised training, they were asked to walk for 30 minutes at home and perform the APA exercises described above.
  Interventions: Other: High intensity exercise
- Sarcopenia and 'usual care' unsupervised exercise (Active Comparator): Participants were required to do 5-12 chair rises and also 30-minutes walking 5 days per week. Upper limb and trunk flexibility exercises were also taught.
  Interventions: Other: Usual care home exercise

INTERVENTIONS:
Other: High intensity exercise — Supervised high-intensity combined-modality exercise was administered to participants in the exercise arm for 3 times per week for 6 months. A post-exercise recovery protein drink (31g whey-based) was given within 15 minutes after each supervised exercise session.
  Arms: Sarcopenia and combined-modality high intensity supervised exercise training
Other: Usual care home exercise — Walking 30 minutes, chair rises and flexibility exercises for trunk and upper extremities 5 days per week
  Arms: Sarcopenia and 'usual care' unsupervised exercise

SUMMARY:
This study examined the effects of combined-modality exercise training (resistance, endurance, flexibility and balance) on muscle mass, muscle function and physical activity in community-dwelling elderly living in Jamaica who had been characterised as having sarcopenia.

DETAILED DESCRIPTION:
Community-dwelling seniors aged 60 years and older were screened for muscle mass and function (grip strength and walk speed) and persons with sarcopenia were identified using the European Working Group on Sarcopenia in Older Persons (EWGSOP) algorithm for case finding (N=1344). Of the 77 seniors with sarcopenia, 38 consented to participate and were randomly allocated to receive 6 months combined-modality high intensity treadmill based exercise and a 'usual care' home exercise programme. A comparison of the effects of treatment assignment on muscle mass, function, fitness, physical activity level and disability was done. Participants in the supervised combined-modality high intensity group were required to attend sessions 3 times per week; participants in the home exercise programme were required to attend 1 supervised session at the start of their 6-month intervention. Outcomes were assessed at baseline and at the end of the 6-month intervention. Data were analysed using standard statistical parametric and non-parametric methods including repeated measures analysis of variance to determine changes in outcomes and regression to establish determinants of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years old,
* independently ambulant, with or without an assistive device
* mentally competent to give informed consent and follow exercise instructions

Exclusion Criteria:

* a history of stroke with residual disability
* a diagnosis of cancer
* neuromuscular disorders
* auto-immune disorders
* dementia
* severe arthritis rendering participation in an exercise programme difficult
* unstable cardiovascular disease which renders exercise unsafe

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Functional endurance | 6 months
  Distance walked in 6 minutes
Disability | 6 months
  Lawton Instrumental Activities of Daily Living scale: minimum score = 0 (low function, dependent); maximum score = 8 (high function, independent). Lower scores indicate a worse outcome.
Lower extremity (LE) functional strength | 6 months
  1-repetition maximum (RM) strength
Accelerometry | 6 months
  weekly energy expenditure
self-selected walk speed | 6 months
  speed in the timed-10-metre walk
Appendicular lean mass index | 6 months
  dual energy x-ray absorptiometry (DEXA) measured appendicular lean mass summed and divided by height squared, expressed in kg/m2
Balance | 6 months
  Berg balance test score: minimum score = 0, maximum score = 56. Lower values indicate worse outcome
Fat-free mass | 6 months
  dual energy x-ray absorptiometry (DEXA) determined: fat mass subtracted from weight, expressed in kg

SECONDARY OUTCOMES:
Depression | 6 months
  Center for Epidemiological Studies-Depression [CES-D] score: minimum score = 0, maximum score = 60, with higher scores indicating more depressive symptoms
Timed-up-and-go | 6 months
  Functional test indicating fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Forrester, PhD, Principal Investigator — UWI Solutions for Developing Countries; Michael Boyne, MD, Principal Investigator — UWI Department of Medicine
Locations (1):
- UWI Solutions for Developing Countries (SODECO), Kingston, KSA, Jamaica